CLINICAL TRIAL: NCT03093207
Title: Evaluation of Omega-3 Polyunsaturated Fatty Acids Plus Low-dose Aspirin Daily Supplementation in Surgical Therapy to Treat Generalized Aggressive Periodontitis: Randomized Controlled Clinical Trial
Brief Title: Omega-3 Fatty Acids Plus Low-dose Aspirin Daily Supplementation in Surgical Therapy to Treat Aggressive Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, PhD Adjunt professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HMT+OFD CFA
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Results first posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Residual Disease; Aggressive Periodontitis
Keywords: Aggressive periodontitis; Aspirin; Omega-3 polyunsaturated fatty acids; Surgical therapy
MeSH Terms: conditions — Neoplasm, Residual; Aggressive Periodontitis | interventions — Docosahexaenoic Acids; Fish Oils; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): In this group (n = 17), patients will take placebo pills and open flap debridement will be performed to treat residual pockets.
  Interventions: Procedure: Open flap debridement; Other: Placebo
- Test Group (Experimental): In this group (n = 17), patients will take 3 g of omega-3 polyunsaturated fatty acids plus 100 mg of aspirin daily supplementation over a period of 180 days and open flap debridement will be performed to treat residual pockets.
  Interventions: Procedure: Open flap debridement; Dietary Supplement: Omega-3 polyunsaturated fatty acids; Drug: Aspirin

INTERVENTIONS:
Procedure: Open flap debridement — Open flap debridement will be performed to decontaminate root surface
  Other Names: Surgical therapy
Other: Placebo — Placebo pills over a period of 180 days
  Arms: Control group
Dietary Supplement: Omega-3 polyunsaturated fatty acids — 3 g of omega-3 polyunsaturated fatty acids daily supplementation over a period of 180 days
  Other Names: Fish oil
  Arms: Test Group
Drug: Aspirin — 100 mg of aspirin daily supplementation over a period of 180 days
  Other Names: acetylsalicylic acid
  Arms: Test Group

SUMMARY:
The aim of this randomized controlled clinical trial of superiority will be to evaluate the effect of 3 g of omega-3 polyunsaturated fatty acids and 100 mg of aspirin daily supplementation over a period of 180 days as adjunct to surgical therapy of residual pockets from patients with generalized aggressive periodontitis. Probing depth, clinical attachment level, gingival index and concentration of microorganisms and cytokines at baseline, 3, and 6 months after the procedure will be evaluated.

DETAILED DESCRIPTION:
The study is designed as a prospective, interventional, parallel, blinded, randomized, controlled clinical trial clinical of superiority, with a 6 month follow-up. The methodology of the present study will follow the standards of CONSORT-STATEMENT 2010 (Moher et al., 2010) and SPIRIT 2013 (Chan et al., 2013) for randomized clinical trials.

Source of data The population will be composed of patients diagnosed with generalized aggressive periodontitis (GAgP) recruited at Institute of Science and Technology - Unesp, in São José dos Campos / SP, who have already undergone non-surgical periodontal treatment and still have pockets with probing depth ≥5 mm and bleeding on probe.

Sample size Sample size calculation was performed using Sealed EnvelopeTM software. For this study, a population of 34 patients will be included. Considering α = 5% and β = 5% (power of 95%) to detect a change of at least 1 mm in clinical attachment level between groups, to a standard deviation of 0.8 mm, 17 patients will be required in each group

Clinical Parameters All clinical parameters will be assessed by a single blinded, trained and calibrated examiner (CFA) before surgical therapy (baseline) and at 3 and 6 months after using a manual probe. Measurements will be done at six sites per tooth (mesiobuccal, buccal, disto-buccal, distolingual, lingual, and mesiolingual) in all teeth, except third molars.

The following clinical parameters will be evaluated: 1) Full-mouth plaque index (PI); 2) Bleeding on probing (BoP); 3) Probing depth (PD): distance from the bottom of sulcus/pocket to gingival margin; 4) Gingival recession (GR): distance from the free gingival margin to cement-enamel junction (CEJ); 5) Clinical attachment level (CAL): distance from bottom of sulcus/pocket to the CEJ. The CEJ will be identified by careful probe on cervical area.

Calibration and Randomization Initially, ten patients with GAgP will be selected. The designated examiner (CFA) will measure CAL and PD in all patients twice within 24 hours, with an interval of ≥ 1 hour between examinations. Then, the measures will be submitted to intraclass correlation test and the examiner will be judged calibrated if reaches 90% agreement.

Patients will be allocated into two groups according to a computer-generated list. The allocation will be implemented by an investigator (NC) who was not directly involved in the examination or treatment procedures.

Selection of sites with residual pockets

After the reevaluation, a residual periodontal pocket with probing depth ≥5 mm and bleeding on probe will be selected from a site not located in furcation region, by chance, to receive one of the following treatments:

* Control group (CG): surgical access for scaling and root planing + placebo pills (n = 17);
* Test group (TG): surgical access for scaling and root planing associated with daily supplementation of 3 g of omega-3 and 100 mg of acetylsalicylic acid for 180 days (n = 17).

Treatment

One hour before surgical therapy, patients will receive a single dose of dexamethasone 4 mg. The packaging of the products will be delivered according to the therapy indicated in the randomization. The administration will begin immediately before the surgical treatment, which will be performed by a single operator (CA), following the sequence:

1. 10 mL of 0.1% chlorhexidine digluconate solution (Periogard®, Colgate Palmolive Ltda - Osasco - SP) will be provided to be chewed by the patient for 1 minute for intraoral disinfection;
2. Antisepsis of the perioral region with sterile gauze soaked in chlorhexidine digluconate solution 0.2%;
3. The patient will receive local injectable anesthesia with mepivacaine 2% with epinephrine 1: 100,000 (Mepivacaína®, DFL - Rio de Janeiro / RJ) through an infiltrative technique;
4. Surgical access will be performed by Kirkland modified surgical technique (Kirland, 1931). With a 15c blade, intrasulcular incisions will be made to the bottom of the pocket / sulcus on buccal, lingual and interproximal surfaces. The incisions will extend into the mesial and distal directions of the affected tooth. The gingival tissue will be detached from the bone to allow exposure of the root surface which will be carefully scaled and plained with periodontal curettes after removal of all granulation tissue. After copious irrigation with saline solution, the flap will be repositioned and maintained by interproximal sutures with Ethicon ® 4-0 silk suture (Ethicon Johnsons do Brasil SA, São José dos Campos - SP).

Postoperative Patients will receive the following postoperative recommendations: do not drink alcoholic beverages; do not touch the surgical wound; Do not brush and floss area for 7 days; Ingest only cold liquid (ice cream, yogurt, juices and gelatin) in the first 24 hours; Mouthwash with 0.12% chlorhexidine digluconate (Periogard®) every 12 hours for 14 days. Dipyrone sodium 500 mg every 4 hours will be prescribed in case of pain. The sutures will be removed after 7 days of surgery.

Microbiological evaluation Subgingival microbiological samples will be collected at the baseline, 3 and 6 months after therapy. The site will be isolated with a sterile cotton roller and supragingival biofilm will be carefully removed with periodontal curettes and a sterile paper will be inserted into the periodontal pocket for 30 s (Hartoth et al., 1999). The sample will be stored in sterile microtubes. The samples will then be lyophilized and sent to the Department of Periodontology at the University of Florida, where the samples will be analyzed.

Evaluation of cytokines For the analysis of immunological changes, crevicular gingival fluid (CGF) will be collected at baseline, 3 and 6 months after treatment. Each site will be isolated with a sterile cotton roller and the supragingival biofilm will be removed. After this, the CGF will be collected with Periopaper strips (Periopaper, Oraflow, Plainview, NY, USA), inserted in the pocket for 15 seconds. The volume of collected fluid will be measured (Periotron 8000, Oraflow). The Periopaper strips will be stored in a sterile tube containing 300μl of phosphate saline (PBS) with 5% Tween-20 and stored in a freezer at -20 ° C until the multiplex test. The level of the following cytokines will be measured in the CGF: interferon (IFN) -γ, interleukins (IL) -10, -1β, -4, -6, -8, tumor necrosis factor (TNF) -α, macrophage inflammatory protein 1α (MIP1α), 1α monocyte chemotactic protein (MCP-1α). The 10-plex high sensitivity kit (Millipore Corporation, Billerica, MA, USA) will be used according to the manufacturer's instruction and analyzed using the MAGpixTM platform (MiraiBio, Alameda, CA, USA). Samples will be analyzed individually (each pocket separately) and the concentrations will be calculated using a standard 5-parameter curve in the Xponet program (Millipore Corporation). The concentration of each marker will be given in pg / ml. All analysis of cytokine concentrations will be done in duplicate.

Statistical analysis Two analyzes will be performed: Per Protocol and Intention-to-treat (Moher, 2010; Gupta, 2011; Day, 2008). For each of them, mean and standard deviation will be calculated in each of the parameters. Full-mouth PI, GI, PD, CAL, and GR will be submitted to the Shapiro-Wilk test to evaluate the distribution of these data, and then subjected to the variance test for both intra- and intra-group comparison. In addition, the number of pockets ≥ 5mm, the frequency of closure of these pockets, the mean reduction in PS and the gain in CAL of these pockets will be assessed before and after the therapy by performing intra- and inter-group analyzes.

The concentration of each cytokine will be analyzed by test of variance for intra and intergroup comparison.

ELIGIBILITY:
Inclusion criteria

* Diagnosis of generalized aggressive periodontitis (Armitage, 1999; American Academy of Periodontology, 2015);
* Have undergone a first approach for periodontal treatment (full-mouth ultrasonic debridement);
* Present at least one residual pocket of probing depth ≥ 5 mm and bleeding on probe not located in furcation region;
* Good general health;
* Agree to participate in the study and sign the informed consent form (TCLE) after explaining the risks and benefits;

Exclusion Criteria

* Systemic problems (cardiovascular alterations, blood dyscrasias, immunodeficiency - ASA III / IV / V) that contraindicate the periodontal procedure;
* Have used antibiotics and anti-inflammatories in the last six months;
* Smoke ≥ 10 cigarettes/day;
* Pregnant or nursing;
* Chronic use of medications that may alter the response of periodontal tissues;
* Indication of antibiotic prophylaxis for dental procedures;
* History of allergic reaction to acetylsalicylic acid, fish or seafood.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2020-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Santamaria, Professor, Principal Investigator — Universidade Estadual Paulista "Julio de Mesquita Filho", ICT/UNESP
Locations (1):
- College of Dentistry - São José dos Campos, Sao Paulo State University, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Sharkawy H, Aboelsaad N, Eliwa M, Darweesh M, Alshahat M, Kantarci A, Hasturk H, Van Dyke TE. Adjunctive treatment of chronic periodontitis with daily dietary supplementation with omega-3 Fatty acids and low-dose aspirin. J Periodontol. 2010 Nov;81(11):1635-43. doi: 10.1902/jop.2010.090628. Epub 2010 Jun 23. PMID 20572767

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: In this group (n = 17), patients received placebo pills and open flap debridement to treat residual pockets.
  Open flap debridement: Open flap debridement was performed to decontaminate root surface
  Placebo: Placebo pills over a period of 180 days
- Test Group: In this group (n = 17), patients received 3 g of omega-3 polyunsaturated fatty acids plus 100 mg of aspirin daily supplementation over a period of 180 days and open flap debridement was performed to treat residual pockets.
  Open flap debridement: Open flap debridement was performed to decontaminate root surface
  Omega-3 polyunsaturated fatty acids: 3 g of omega-3 polyunsaturated fatty acids daily supplementation over a period of 180 days
  Aspirin: 100 mg of aspirin daily supplementation over a period of 180 days
Period: Overall Study
Arm/Group | Control Group | Test Group
Started | 17 | 17
Completed | 17 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Test Group | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 17 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.06 (5.13) | 34.17 (4.9) | 33.61 (5.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Patients were recruited at São José dos Campos, São Paulo, Brazil
  participants
    Brazil | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Clinical Attachment Level at Baseline, 3 Months and 6 Months
Description: Evaluate the difference between baseline and 6 months CAL measures. CAL: distance from bottom of sulcus/pocket to the cement-enamel junction (CEJ). The CEJ will be identified by careful probe on cervical area.
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Error); unit: mm
Units Other Than Participants: Pockets treated with surgery
Groups:
- Control Group: In this group (n = 17), patients received placebo pills over a period of 180 days and open flap debridement was performed to treat residual pockets.
  Open flap debridement: Open flap debridement was performed to decontaminate root surface
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 17 | 17
Number analyzed (Pockets treated with surgery) | 17 | 17
mm
  Baseline | 5.5 (0.25) | 5.29 (0.16)
  3 months | 4.64 (0.29) | 4.73 (0.28)
  6 months | 4.64 (0.22) | 4.97 (0.25)

2. Secondary Outcome: Probing Depth at Baseline, 3 Months and 6 Months
Description: Evaluate the difference between baseline and 6 months PB measures. PB: distance from the bottom of sulcus/pocket to gingival margin.
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Pockets treated with surgery
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 17 | 17
Number analyzed (Pockets treated with surgery) | 17 | 17
mm
  Baseline | 5.17 (0.2) | 5.14 (0.14)
  3 months | 4.08 (0.21) | 3.76 (0.2)
  6 months | 4 (0.15) | 3.94 (0.2)

3. Secondary Outcome: Percentage of Sites With Bleeding on Probe at Baseline, 3 Months and 6 Months
Description: Evaluate the difference between baseline and 6 months BoP measures. BoP: bleeding that is induced by gentle probing of the sulcus/pocket.
Time Frame: Baseline, 3 and 6 months
Measure: Number; unit: percentage of sites with BoP
Units Other Than Participants: Pockets treated with surgery
Arm/Group | Test Group | Control Group
Number analyzed (Participants) | 17 | 17
Number analyzed (Pockets treated with surgery) | 17 | 17
percentage of sites with BoP
  Baseline | 100 | 100
  3 months | 76.47 | 100
  6 months | 64.7 | 64.7

ADVERSE EVENTS:
Time Frame: During the 6 months post-treatment
Arm/Group | Control Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=17) | Test Group (N=17)
Stomachache (Gastrointestinal disorders) | 0 (0) | 0 (0)
Internal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT03093207/Prot_SAP_000.pdf